CLINICAL TRIAL: NCT07035093
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Retatrutide Once Weekly in Participants Who Have Obesity or Overweight and Chronic Low Back Pain
Brief Title: A Study of Retatrutide (LY3437943) in Participants Who Have Obesity or Overweight and Chronic Low Back Pain
Acronym: TRIUMPH-7
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27278; J1I-MC-GZQD (Other: Eli Lilly and Company); 2024-517431-43-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-28; First posted 2025-06-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight; Chronic Low Back Pain (CLBP)
Keywords: Axial Predominant Low Back Pain
MeSH Terms: conditions — Obesity; Overweight | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Retatrutide (Experimental): Participants will receive Retatrutide subcutaneously (SC)
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive Placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of retatrutide in relieving chronic low back pain in participants who have obesity or overweight. Participation in the study will last about 80 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of axial-predominant low back pain
* Have pain that is restricted to the low back or with a referral pattern limited to the proximal legs
* Have a body mass index (BMI) ≥27 kilograms per square meter (kg/m2) at screening
* Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* Have a non-axial origin low back pain
* Have had botulinum or steroid injections to the spine within 1 year of screening
* Have had trigger point injection to the spine within 6 months of screening
* Have a self-reported change in body weight >5 kilograms (kg) (11 pounds) within 90 days prior to screening
* Have been taking drugs to promote body weight reduction, including over-the-counter medications, within 90 days prior to screening
* Have a prior or planned surgical treatment for obesity
* Have Type 1 Diabetes, Type 2 Diabetes, or any other type of diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain Intensity Per Numeric Rating Scale | Baseline, up to 72 weeks
Percent Change from Baseline in Body Weight | Baseline, up to 72 weeks

SECONDARY OUTCOMES:
Number of Participants with Reduction in Pain Intensity Per Numeric Rating Scale | Baseline, up to 72 weeks
Number of Participants with Reduction in Body Weight | Baseline, up to 72 weeks
Change in Physical Function as Measured by Patient-Reported Outcomes Measurement Information Systems (PROMIS) | Baseline, up to 72 weeks
Change in Pain Interference as Measured by PROMIS | Baseline, up to 72 weeks
Change in Sleep as Measured by PROMIS | Baseline, up to 72 weeks
Change in Patient Reported Health Outcomes as Measured by Medical Outcomes Study 36-item Short Form Health Survey version 2 (SF-36v2) | Baseline, up to 72 weeks
Change in Waist Circumference | Baseline, up to 72 weeks
Change in Biomarkers of Inflammation as Measured by Blood Test | Baseline, up to 72 weeks
Change in Blood Pressure | Baseline, up to 72 weeks
Change in Glycemic Control | Baseline, up to 72 weeks
Percent Change in Total Cholesterol | Baseline, up to 72 weeks
Percent Change in Urine Albumin-to-Creatinine Ratio (UACR) | Baseline, up to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (47):
- United States (25):
  - MD First Research - Chandler, Chandler, Arizona
  - Tucson Orthopaedic Institute - North Wyatt Drive, Tucson, Arizona
  - Ark Clinical Research - Fountain Valley, Fountain Valley, California
  - St Joseph Heritage Healthcare, Fullerton, California
  - Clinical Research Institute, Los Angeles, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - K2 Medical Research - Daytona Beach, Daytona Beach, Florida
  - Flourish Research - Miami, LLC, Miami, Florida
  - IMA Clinical Research St. Petersburg, St. Petersburg, Florida
  - Care Access - Tampa, Tampa, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Conquest Research, Winter Park, Florida
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Care Access - Lake Charles (Bayou Pines), Lake Charles, Louisiana
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Clinvest Headlands Llc, Springfield, Missouri
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - New Phase Research and Development, Knoxville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Mercy Family Clinic, Dallas, Texas
  - Houston Research Institute, Houston, Texas
  - Sovah Clinical Research-River District, Danville, Virginia
- Argentina (9):
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - CIPREC, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - Centro Rosarino de Investigaciones Clinicas (CRICs), Rosario
  - Instituto Médico Catamarca IMEC, Rosario
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
- Canada (5):
  - Aggarwal and Associates Limited, Brampton
  - Winterberry Research Inc., Hamilton
  - Bluewater Clinical Research Group Inc., Sarnia
  - Care Access - Cape Breton, Sydney
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto
- Mexico (7):
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara
  - Centro de Investigación Clinica Chapultepec, Mexico City
  - Kohler & Milstein Research S.A. De C.V., Mérida
  - IMED Internal Medicine Clin Trials, Monterrey
  - Centro de investigación y control metabólico, Monterrey
  - Arké SMO S.A de C.V, Veracruz
- Podlaskie Centrum Psychogeriatrii, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Retatrutide (LY3437943) in Participants Who Have Obesity or Overweight and Chronic Low Back Pain (TRIUMPH-7) — https://trials.lilly.com/en-US/trial/620575